CLINICAL TRIAL: NCT05766930
Title: A Novel Electrolyzed Water Spray Reduces the Itching Scores of Patients With Genital Itching: A Clinical Study
Brief Title: The Novel Electrolyzed Water Spray Treatment the Genital Itching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jia19951210
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-02

CONDITIONS: Genital Inflammation; Itching
Keywords: Electrolyzed water device; Hydroxyl radical; Tap water; Spray; Genital itching
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: An open label, single arm and before and after treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The genital itching and one treatment (Experimental): Participants with itching genitalia will receive one treatment with the device and complete the questionnaire.
  Interventions: Device: The novel electrolyzed water spray

INTERVENTIONS:
Device: The novel electrolyzed water spray — Study staff will use the novel electrolyzed water spray device and spray for approximately 2-4 minutes on the participant's diseased area until half a bottle (20-40ml) of water is used. The patients use electrolyzed water to treat the diseased area, two times a day, for 5 days. The trial consists of 5 study visits (day 1-day 5). The relief genital itching evaluation and adverse event assessments will be performed at each visit. Safety analysis will be assessed based on the reports of adverse events during the study.

SUMMARY:
The purpose of this study is to test whether spraying the genitalia of patients by use of the novel electrolyzed water spray will produce improvement in the condition of genitalia itching.

DETAILED DESCRIPTION:
In this study, water inculding tap water,pure water and salt water, and an apparatus for producing electrolyzed water (https://www.deposon.com.cn; https://www.deposon.com）were used to generate an electrolyzed water mist spray or spray. This instantly generated electrolyzed water mist spray or spray has oxidation-reduction potential (ORP) ≥1200mv,and contains non-specific total oxidation capacity which equals to 0.28±0.10ppm,0.06±0.04ppm and 3.92±0.39ppm of desolved ozone. This instantly generated electrolyzed water mist spray or spray does not release detectable ≥0.1mg/m3 of gaseous ozone. This instantly generated electrolyzed water mist spray or spray has pH 8.4±0.4 and releases negative air ion.The apparatus for producing electrolyzed water has a positive electrode which is covered by a conductive diamond material (Patent# CN215308550U).

This is an open-label, single-arm, and before and after treatment comparison study. This study uses this novel electrolyzed water device and the water spray to treat genital itching.

ELIGIBILITY:
Inclusion Criteria:

Patients with genital itching.

Exclusion Criteria:

Severe genital itching. 80 years or older.

Ages: 40 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
An itching scale made by modifying a pain scale (NPRS) | 5 days
  This Score is based on descriptions of the itching that patients rate 0-10 to assess the condition of their genitalia with itching. A higher score means a worse outcome. 0 means "no itching " and 10 means "the most itching".

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: until publication of this clinical study and international patent granted